CLINICAL TRIAL: NCT02493595
Title: Post-CE Marking Continuing Evaluation of Multi-Static Microwave Imaging of the Female Breast in Controlled Trial to Identify Optimum Use of the MARIA Platform in the Clinical Workflow
Brief Title: Synthetic Aperture Radar Detection of Breast Tumours
Acronym: MARIA
Status: Completed | Type: Observational
Sponsor: Micrima, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: M5-1
Record Dates: First submitted 2015-04-14; First posted 2015-07-09 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Mammogram Scheduled

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer: Patients attending One-stop Symptomatic Breast Care clinics with suspicion of a breast lesion in one or both breasts.

SUMMARY:
The study will seek to understand the effective use of a novel Microwave Radar Breast Imaging System in a Symptomatic Breast Care Clinic. The MARIA Imaging system uses low level non--ionising radiation (radio wave) signals to scan the breast tissue volume and to provide a visual image of areas of varying tissue permittivity value within the volume. These areas of varying permittivity can be shown as a two or three dimensional image and used in conjunction with the X-Ray mammogram and ultrasound scans to provide another level of diagnosis to the radiologist.The system works equally well in both dense and lucent breast types and can in particular provide insight into the diagnosis in dense tissue cases. The trial will accept symptomatic cases with suspected cancer, cysts or fibroadenoma.

The trial will use the images produced by the MARIA system and compare them to the images obtained using X-Ray mammography. The results of the comparison will be assessed to understand the effectiveness of the MARIA image in assisting with the identification and location of suspected lesions for further specific analysis using Ultrasound/Biopsy.

DETAILED DESCRIPTION:
A potential participant will be asked by the breast care clinician if she would be interested in participating in a new form of breast scanning trial; if agrees to consider is given an patient information sheet and a brief explanation. After the initial consultation and either whilst waiting for, or just after the mammogram, will be approached by the researcher (who is a healthcare professional) to ask if she would like to take part.

Equipment is shown and procedure explained, and if in agreement will be required to sign four copies of the consent form. The patient will be asked to remove top clothing and lie prone on a specifically designed couch that allows one breast to sit in a ceramic cup containing a small amount of contact liquid. The cup position is adjusted to get best fit which is tested with short trial scans taking a few seconds each. Once satisfactory the subject is asked to keep as still as possible for a 25 second scan. The radiowave array is rotated a few degrees and the scan repeated up to four times.

The scanning procedure takes about 3 to 5 minutes in total, but with questions, consent, explanation and dressing the total visit time is about 20 to 25 minutes. The patient is returned to the breast care clinic to continue with investigation and management. Personal details collected at the time are the subject's age, menopausal status and breast (bra) size. Details retrieved from the hospital record system later are the fully anonymised mammogram, ultrasound scan and cytology/histology reports if available. No other intervention is needed.

ELIGIBILITY:
Inclusion Criteria:

* Referred for diagnosis because of a reported symptom of breast disease
* No previous treatment or biopsy
* Breast size 32A to breast size 42DD
* Able to lie prone on a couch for 10 minutes
* Able to remain reasonably still for 2 minutes

Exclusion Criteria:

* Breast implants
* Recent Biopsy
* Extremely small or extremely large breasts
* Presence of metal or blood lesion (haematoma)
* Breathlessness or severe arthritis

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female Patients with suspicion of breast lesions attending One-Stop Breast Care diagnostic clinics
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Radio-Wave imaging in the diagnostic breast care clinic | Duration of the Study, 6 month interval progress assessment
  The research will seek to measure the added value of a radiowave imaging procedure in a diagnostic breast care clinic in improving accuracy of diagnostic outcomes. In particular it will evaluate the ability of radiowave imaging in the younger patient to demonstrate the presence of lesions in tissue which is dense. As a nonionizing radiation it also has potential to be the bulk imaging method of choice in women under 40 who would only be offered a mammogram where the risk benefit justified it, i.e. with a probability of malignancy.

SECONDARY OUTCOMES:
Comparison of radio wave image sensitivity in Dense Tissue BIRADS c and d as compared to X-Ray Mammography | Study result assessed every 6 months
  MARIA image sensitivity will be assessed separately for patients with Higher density breast tissue

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Shere, M.R.C.S, Principal Investigator — North Bristol NHS Trust, United Kingdom
Locations (1):
- North Bristol Trust NHS Breast Care Clinic, Bristol, United Kingdom